CLINICAL TRIAL: NCT03322358
Title: Chronic Sleep Deprivation Among the Poor: A Lab-in-the-field Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Institute for Financial Management and Research (Other); Abdul Latif Jameel Poverty Action Lab (Other); Government of Tamil Nadu, India (Other)
Responsible Party: Principal Investigator, Heather Schofield, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 14-2294
Record Dates: First submitted 2017-10-12; First posted 2017-10-26 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-11

CONDITIONS: Blood Pressure; Depression
MeSH Terms: conditions — Depression | interventions — N-(4-aminophenethyl)spiroperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (No Intervention): No changes to normal sleep habits.
- Naps only (Experimental): After a baseline period, participants in this condition will be provided with the opportunity to nap in a quiet comfortable "nap cabin" in the study office for 30 minutes each afternoon on all work days.
  Interventions: Other: Naps
- Home sleep aids only (Experimental): After a baseline period, participants in this condition will be provided with a set of home sleep aids (e.g. earplugs, eyeshades, a basic mattress, sheets, and pillow, etc) to take home with them if they wish. These sleep aids and their proper use are described to the participants and they are encouraged to use them if they find them helpful.
  Interventions: Device: Home sleep aids
- Home sleep aids + Sleep incentives (Experimental): After a baseline period, participants in this condition will be provided with a set of home sleep aids (e.g. earplugs, eyeshades, a basic mattress, sheets, and pillow, etc) to take home with them if they wish. These sleep aids and their proper use are described to the participants and they are encouraged to use them if they find them helpful. In addition, they will be given a small payment for each additional minute of sleep over their mean nighttime sleep in the baseline period.
  Interventions: Device: Home sleep aids; Other: Sleep incentives
- Naps + Home sleep aids (Experimental): After a baseline period, participants in this condition will be provided with: 1) the opportunity to nap in a quiet comfortable "nap cabin" in the study office for 30 minutes each afternoon on all work days, 2) a set of home sleep aids (e.g. earplugs, eyeshades, a basic mattress, sheets, and pillow, etc) to take home with them if they wish. These sleep aids and their proper use are described to the participants and they are encouraged to use them if they find them helpful.
  Interventions: Other: Naps; Device: Home sleep aids
- Naps + Home sleep aids + Sleep incentives (Experimental): After a baseline period, participants in this condition will be provided with: 1) the opportunity to nap in a quiet comfortable "nap cabin" in the study office for 30 minutes each afternoon on all work days, 2) a set of home sleep aids (e.g. earplugs, eyeshades, a basic mattress, sheets, and pillow, etc) to take home with them if they wish, and 3) a small payment for each additional minute of sleep over their mean nighttime sleep in the baseline period. The sleep aids and their proper use are described to the participants and they are encouraged to use them if they find them helpful.
  Interventions: Other: Naps; Device: Home sleep aids; Other: Sleep incentives

INTERVENTIONS:
Other: Naps — After a baseline period, participants in this condition will be provided with the opportunity to nap in a quiet comfortable "nap cabin" in the study office for 30 minutes each afternoon on all work days.
  Arms: Naps + Home sleep aids; Naps + Home sleep aids + Sleep incentives; Naps only
Device: Home sleep aids — After a baseline period, participants in this condition will be provided with a set of home sleep aids (e.g. earplugs, eyeshades, a basic mattress, sheets, and pillow, etc) to take home with them if they wish. These sleep aids and their proper use are described to the participants and they are encouraged to use them if they find them helpful.
  Arms: Home sleep aids + Sleep incentives; Home sleep aids only; Naps + Home sleep aids; Naps + Home sleep aids + Sleep incentives
Other: Sleep incentives — After a baseline period, participants in this condition will be provided with a small payment for each additional minute of sleep over their mean nighttime sleep in the baseline period.
  Arms: Home sleep aids + Sleep incentives; Naps + Home sleep aids + Sleep incentives

SUMMARY:
A large body of medical research has shown that sleep deprivation adversely affects outcomes ranging from cognitive function to pain sensitivity and cardiovascular function. Much of this evidence comes from sleep labs in the developed world, where sleep can be carefully manipulated, and short-run physiological and cognitive outcomes precisely measured. In contrast, there is much less knowledge about how sleep deprivation affects the health of individuals in the developing world, coming from a lack of studies outside the lab and over longer periods. This project aims to fill this gap. The investigators will implement a randomized controlled trial (RCT) with 450 low-income adults in Chennai, India, providing the first objective measurement of sleep in a developing country. The investigators will also evaluate scalable interventions to improve the sleep of poor adults, such as providing home sleep-aid devices and a comfortable space for a 30-minute afternoon nap at the participants' work site. Finally, the study aims to assess the impact of improved sleep on health, with a primary focus on cardiovascular health and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Unemployed and underemployed adult men and women of working age (see previous age limit) who have worked less than 5 days per week over the last month and earned less than Rs. 700 per day over that same period.
* Participants must live in Government board house or in a house with some kind of roof that protect the sleep aids from rain, such as a concrete or a metal or a Tarpaulin, ... roof.
* Have limited experience with typing, and limited knowledge of English.
* Participants need to speak Tamil, the local language, to be able to write numbers and to be able to commit easily to the office.

Exclusion Criteria:

* Participants who cannot commit to come to the office for the duration of the whole study.
* Participants who own more than three of the sleep aids that we provide in our sleep kit.
* Participants who have previously participated in the sleep study.
* Participants who have children younger than three years old.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 452 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Rao, PhD, Principal Investigator — Harvard University; Frank Schilbach, PhD, Principal Investigator — Massachusetts Institute of Technology; Margaret McConnell, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (2):
- India (2):
  - Institute for Financial Management and Research, Chennai, Tamil Nadu
  - J-PAL South Asia, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Yes
We will make the de-identified data available upon request after publication.
Supporting Information: Study Protocol, ICF
Time Frame: After publication.

REFERENCES:
- [Result] Bessone P, Rao G, Schilbach F, Schofield H, Toma M. The Economic Consequences of Increasing Sleep Among the Urban Poor. Q J Econ. 2021 Apr 8;136(3):1887-1941. doi: 10.1093/qje/qjab013. eCollection 2021 Aug. PMID 34220361
- Available data/document: Individual Participant Data Set — https://www.sleepdata.org/datasets/urbanpoor

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Started | 77 | 75 | 75 | 74 | 75 | 76
Completed | 77 | 75 | 75 | 74 | 75 | 76
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives | Total
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76 | 452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 77 | 75 | 75 | 74 | 75 | 76 | 452
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.91 (0.86) | 35.77 (0.89) | 35.04 (0.80) | 33.82 (0.74) | 35.52 (0.85) | 33.62 (0.83) | 34.95 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 48 | 47 | 48 | 56 | 299
  Male | 25 | 27 | 27 | 27 | 27 | 20 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 77 | 75 | 75 | 74 | 75 | 76 | 452
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 77 | 75 | 75 | 74 | 75 | 76 | 452
Region of Enrollment [Number; unit: participants]
  India | 77 | 75 | 75 | 74 | 75 | 76 | 452
Hours of sleep/24 hours [Mean (Standard Deviation); unit: Hours of sleep/24 hours] — This outcome measures the average number of hours of sleep for each participant per day during the baseline period, i.e. before the treatment starts. Sleep is measured using actigraphs. Total 24 hour sleep is the number of hours of night sleep plus the number of hours of nap sleep.
  Hours of sleep/24 hours | 5.509 (1.261) | 5.584 (1.204) | 5.588 (1.186) | 5.640 (1.118) | 5.542 (1.291) | 5.567 (1.144) | 5.581 (1.197)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Per 24 Hours
Description: Sleep is measured via actigraph. 24 hour sleep is the sum of night sleep and nap sleep.
Time Frame: Actigraphs are worn consistently throughout the study. The sleep per 24 hour period outcome is then measured every day through study completion, which is 28 business days (as well as intervening holidays and Sundays) for each participant.
Measure: Mean (Standard Deviation); unit: Hours of sleep/24 hours
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Hours of sleep/24 hours | 5.61 (1.200) | 5.81 (1.259) | 5.99 (1.239) | 6.23 (1.312) | 6.08 (1.305) | 6.35 (1.208)

2. Secondary Outcome: Blood Pressure
Description: Systolic, Diastolic. The outcome measurements reported here are those captured after the baseline period (starting on day 9). Each measure is first winsorized at the 5% level and standardized using control group data, to mean 0 and standard deviation 1. The measure is then multiplied by -1 such that higher values represent improvements in health. In order to analyze these outcomes jointly, this measure is next averaged to obtain an overall measure and standardized again. The mean is taken across all participant observations within a group regardless of the time after the baseline period. There are no clinically relevant values and the measure has no max and min.
Time Frame: From date of entering the study through completion of the study after 28 business days, blood pressure is measured once every block of three business days. The date of measurement is randomized within each block between the first, second, and third day.
Measure: Mean (Standard Deviation); unit: Blood pressure index
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Blood pressure index | 0.000 (1.000) | 0.135 (0.891) | 0.110 (0.981) | 0.071 (0.950) | 0.027 (1.025) | 0.178 (0.902)

3. Secondary Outcome: Depression
Description: The investigators measure depression using a scale defined by the Patient Health Questionnaire (PHQ), which is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. Each criteria is scored from "0" (not at all, a better outcome) to "3" (nearly every day, a worse outcome). Scores on each question are summed, defining depression severity. The outcome measure was the total summed score captured at endline (day 28). The outcome is thus measured on a scale from 0 to 27, where 0 represents the best outcome and 27 represents the worst outcome.
Time Frame: Depression is measured once in the baseline on the first day of the study and a second time in the endline, which takes place on the last day of the study, 28 business days after the first day in the study for the participant.
Measure: Mean (Standard Deviation); unit: Score on 0-27 scale
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Score on 0-27 scale | 5.208 (5.131) | 4.676 (4.726) | 5.851 (5.529) | 5.095 (5.113) | 5.608 (5.226) | 5.147 (5.339)

4. Secondary Outcome: Number of Days of Illness in Past Week
Description: Illness is measured as the number of days of illness (e.g. cough, fever) in the past week. The outcome measure is the number of days of illness in the past week self-reported at endline (day 28).
Time Frame: Illness is measured once in the baseline on the first day of the study and a second time in the endline, which takes place on the last day of the study, 28 business days after the first day in the study for the participant.
Measure: Mean (Standard Deviation); unit: Days of illness in the past week
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Days of illness in the past week | 2.08 (2.448) | 1.732 (1.836) | 1.973 (2.560) | 2.041 (2.556) | 2.351 (2.550) | 1.853 (2.228)

5. Secondary Outcome: Inhibitory Control
Description: Hearts and flowers test -- The outcome used is the payment for the task which is a linear combination of the participant's accuracy (percent correct) and reaction time (measured in milliseconds). Specifically, the payment for this task is determined by the formula: 1.5 * ((percent correct - 0.84) / 0.2 - (reaction time - 526.5) / 95.2) + 15. The outcome measure is the average of the measures collected for each individual after the baseline period (starting on day 9).
Time Frame: From date of entering the study through completion of the study after 28 business days, the inhibitory control is measured once every two business days (which of the two is randomly assigned).
Measure: Mean (Standard Deviation); unit: Indian Rupees
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Indian Rupees | 14.982 (1.371) | 14.957 (1.328) | 15.078 (1.213) | 14.982 (1.086) | 15.039 (1.338) | 15.103 (1.301)

6. Secondary Outcome: Memory
Description: Corsi block span - The investigators' measure of memory is the longest correct sequence of blocks lighting in a random order that a participant can reproduce. The range is from a minimum of 0 (worst performance) to a maximum of 9 (best performance). The outcome reported for this task is the participant's payment from the task, which is computed based on their longest span as well as baseline data: 2.29*(maximum span - 5.3) / 1.17 + 13. The outcome measure is the average of the measures collected for each individual after the baseline period (starting on day 9).
Time Frame: From date of entering the study through completion of the study after 28 business days, memory is measured once every two business days (which of the two is randomly assigned).
Measure: Mean (Standard Deviation); unit: Indian Rupees
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Indian Rupees | 14.643 (2.675) | 14.834 (2.519) | 14.931 (2.499) | 14.483 (2.384) | 14.609 (2.796) | 14.645 (2.608)

7. Secondary Outcome: Attention
Description: Psychomotor Vigilance Task (PVT) - The outcome is payment for the task which was a predetermined linear combination of the inverse reaction time, the number of false positives (response when they participant should not have responded), and the number of lapses (reaction time >500ms). Specifically, the payment was determined by the formula: (inverse reaction time - 3.5)/0.42 - (0.5*(number of false positives-4.7)/6.14) - (0.5*(number of lapses-1.3)/2.58) + 15. Higher payments indicate better performance. Although the theoretical minimum possible score is negative infinity, in practice, the minimum possible payment was censored at zero. The maximum theoretical payment is undefined. The payment reflects overall performance. The outcome measure is the average of the measures collected for each individual after the baseline period (starting on day 9).
Time Frame: From date of entering the study through completion of the study after 28 business days, attention is measured once every two business days (which of the two is randomly assigned).
Measure: Mean (Standard Deviation); unit: Indian Rupees
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Indian Rupees | 13.001 (1.568) | 13.338 (1.418) | 13.024 (1.569) | 13.005 (1.518) | 13.174 (1.589) | 13.150 (1.495)

8. Secondary Outcome: Self-reported Pain
Description: The investigators use a simple scale of 0 (no pain) to 10 (the worst pain imaginable) for the participant to rate their pain intensity. The outcome measure was the self-reported pain intensity captured at endline (day 28).
Time Frame: Pain is measured once in the baseline on the first day of the study and a second time in the endline, which takes place on the last day of the study, 28 days after the first day in the study for the participant.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Score on a scale | 2.740 (2.721) | 3.070 (2.276) | 2.095 (2.517) | 2.838 (2.477) | 2.608 (2.520) | 2.800 (2.568)

9. Secondary Outcome: Physical Fitness
Description: The outcome measure is the number of kilometers participants can cover on a stationary exercise cycle over a period of 30 minutes, as reported on the display of the exercise cycle.The cycle was set to the same level of resistance for all participants.
Time Frame: Physical fitness is measured only once in the endline, which takes place on the last day of the study, 28 business days after the first day in the study for the participant.
Measure: Mean (Standard Deviation); unit: km
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
km | 3.717 (1.626) | 3.857 (1.357) | 3.941 (1.924) | 3.934 (2.157) | 3.697 (1.446) | 3.571 (1.384)

10. Secondary Outcome: Activities of Daily Living
Description: The investigators use survey questions taken from the commonly used SF-36 Health survey asking participants how much their health has limited them in a certain number of activities. The possible answers range from "they did not limit you at all" (0, the best outcome) to "limited you a lot" (3, the worst outcome). The final scale, which is the sum of the answers, goes from 0 for people who are not limited at all in their daily life by their health to 36 for people who are substantially limited in their daily life by their health. The outcome measure is the 0-36 scale captured at endline (day 28).
Time Frame: Activities of daily living are measured once in the baseline on the first day of the study and a second time in the endline, which takes place on the last day of the study, 28 business days after the first day in the study for the participant.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Score on a scale | 8.961 (7.378) | 7.52 (6.795) | 7.8 (7.674) | 7.486 (7.323) | 7.36 (6.060) | 7.553 (7.430)

11. Secondary Outcome: Subjective Well-being
Description: The measure of the outcome is based on two survey questions taken from Gallup Survey. In the first question, participants are asked to state a number from 0 to 10, with 0 being a feeling that the participant has the worst possible life while 10 is a feeling that the participant has the best possible life. In the second question, participants are asked to state a number from 0 to 10, with 0 being a feeling that the participant is dissatisfied with life as a whole and 10 being a feeling that the participant is satisfied with life as a whole. The final scale, generated by summing the individual items, is then from 0 for highly dissatisfied people to 20 for highly satisfied people. The outcome measure is the 0-20 scale captured at endline (day 28).
Time Frame: Subjective well-being is measured once in the baseline on the first day of the study and a second time in the endline, which takes place on the last day of the study, 28 business days after the first day in the study for the participant.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Score on a scale | 11.554 (4.78) | 12.521 (4.004) | 11.906 (4.588) | 11.919 (4.336) | 12.757 (4.132) | 12.199 (4.489)

12. Secondary Outcome: Happiness
Description: The investigators use a question adapted from a Gallup poll and from the SF-36 survey by RAND that ask participants to rate their happiness on the present day from "Not at all happy" (0, the worst outcome) to "very happy" (4, the best outcome). The outcome measure is the average of the measures collected for each individual after the baseline period (starting on day 9)
Time Frame: Happiness is measured in the baseline on the first day of the study, randomly once every block of three business days during the study, and a last time in the endline, on the last day of the study, 28 business days after the participant's first day.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
Number analyzed (Participants) | 77 | 75 | 75 | 74 | 75 | 76
Score on a scale | 2.455 (0.758) | 2.517 (0.768) | 2.421 (0.754) | 2.440 (0.725) | 2.580 (0.676) | 2.502 (0.783)

ADVERSE EVENTS:
Time Frame: 4 weeks per participant (the duration of each participant's engagement with the study)
Description: Death and serious adverse events follow standard definitions. Participants were seen daily at the study office and PIs continuously monitored for the occurrence of such events with the help of local project leaders.
Arm/Group | Control | Naps Only | Home Sleep Aids Only | Home Sleep Aids + Sleep Incentives | Naps + Home Sleep Aids | Naps + Home Sleep Aids + Sleep Incentives
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/75 | 0/75 | 0/74 | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/75 | 0/75 | 0/74 | 0/75 | 0/76
Other Adverse Events (participants affected / at risk) | 0/77 | 0/75 | 0/75 | 0/74 | 0/75 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03322358/Prot_001.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03322358/SAP_002.pdf
  • Informed Consent Form (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03322358/ICF_000.pdf